CLINICAL TRIAL: NCT02152605
Title: A 12 Week, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy of Umeclidinium/Vilanterol 62.5/25mcg in Subjects With COPD
Brief Title: A Phase IIIb Study to Evaluate the Efficacy of Umeclidinium/Vilanterol (UMEC/VI) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201211
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: SGRQ; vilanterol; long-acting beta2-agonist; long-acting muscarinic antagonist; COPD; umeclidinium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium/Vilanterol 62.5/25 mcg once daily (Experimental): The subjects will receive UMEC/VI 62.5/25 mcg, administered as one inhalation once-daily in the morning via a dry powder inhaler (DPI)
  Interventions: Drug: UMEC/VI
- Placebo once daily (Placebo Comparator): The subjects will receive placebo, administered as one inhalation once-daily in the morning via a DPI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UMEC/VI — Dry white powder delivered via DPI (2 strips with 30 blisters each, first containing UMEC 62.5 mcg per blister and second containing VI 25 mcg per blister), administered as one inhalation of UMEC/VI 62.5/25 mcg
  Arms: Umeclidinium/Vilanterol 62.5/25 mcg once daily
Drug: Placebo — Dry white powder delivered via DPI (2 strips with 30 blisters each, both containing lactose with magnesium stearate), administered as one inhalation of placebo
  Arms: Placebo once daily

SUMMARY:
This study is a 12-week, multicenter, randomized, double blind, parallel group, placebo-controlled study.

The purpose of this study is to replicate the therapeutic benefit of UMEC/VI 62.5/25 microgram (mcg) on health-related quality of life as reflected by St. George's Respiratory Questionnaire (SGRQ) scores and symptoms as reflected by rescue medication use observed in the 6 month placebo controlled study (DB2113373). Lung function will be assessed as it provides an objective measure to support the subjective patient reported outcomes of SGRQ and rescue medication use. The study is intended to provide additional evidence to support the use of UMEC/VI for the maintenance treatment of COPD Approximately 496 subjects will be randomized from approximately 62 centers in order to ensure 422 subjects complete 12 weeks of treatment. Eligible subjects will be randomized to UMEC/VI 62.5/25mcg or placebo in a 1:1 ratio. All treatments will be administered once-daily in the morning via a Dry Powder Inhaler (DPI).

There will be a total of 5 clinic visits. The total duration of study participation will be approximately 15 weeks. All subjects will be provided with albuterol/salbutamol to use as needed for the relief of COPD symptoms throughout the run-in and double-blind treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: 40 years of age or older at Visit 1.
* Gender: Male and female subjects are eligible to participate in the study.
* A female subject is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile (For example [e.g.] age appropriate, >45 years, in the absence of hormone replacement therapy; or child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label, if appropriate, and the instructions of the physician for the duration of the study screening to follow-up contact): abstinence; oral contraceptive (either combined or progestogen alone); injectable progestogen; implants of levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label; male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study (this male is the sole partner for that subject); and double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g. 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack-year history.
* Severity of Disease: A pre and post-albuterol/salbutamol FEV1/ Forced Vital Capacity (FVC) ratio of <0.70 and a post-albuterol/salbutamol FEV1 of <=70% of predicted normal values calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations at Visit 1.
* Dyspnea: A score of >=2 on the Modified Medical Research Council (mMRC) Dyspnea Scale at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: Any subject who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any subject who has any condition (e.g. neurological condition) that is likely to affect respiratory function should not be included in the study.
* Severe Hepatic Impairment: Patients with severe hepatic impairment (Child-Pugh class C) should be excluded unless, in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Unstable or life threatening cardiac disease: UMEC/VI should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: myocardial infarction or unstable angina in the last 6 months; unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV heart failure.
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, sympathomimetic, lactose/milk protein or magnesium stearate.
* Antimuscarinic effects: Subjects with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction should only be included if, in the opinion of the study physician, the benefit outweighs the risk.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead Electrocardiogram (ECG): Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. Subjects with the following abnormalities are excluded from participation in the study: Atrial fibrillation with rapid ventricular rate >120 beats per minute (bpm); Sustained or non-sustained ventricular tachycardia; Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted).
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Interactions: Concomitant administration with beta-blockers and strong Cytochrome P450 3A4 (CYP3A4) inhibitors is only permitted if, in the Investigator's opinion, the likely benefit outweighs the potential risk.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids (12 weeks), systemic, oral or parenteral corticosteroids (6 weeks), antibiotics (for lower respiratory tract infection) (6 weeks), Long acting Beta-Agonist (LABA)/ Inhaled Corticosteroid (ICS) combination products if LABA/ICS therapy is discontinued completely (30 days), LABA/ICS combination products only if discontinuing LABA/ICS therapy and switching to ICS monotherapy (48 hours for salmeterol or formoterol component and 14 days for vilanterol component), ICS (dose >1000 mcg/day of fluticasone propionate or equivalent) (30 days), Initiation or discontinuation of ICS use (30 days), Phosphodiesterase 4 (PDE4) Inhibitor (roflumilast) (14 days), Inhaled long acting beta2 agonists (48 hours for salmeterol, formoterol, 14 days for olodaterol, indacaterol), Long-acting muscarinic antagonists (tiotropium, aclidinium, glycopyrronium, umeclidinium) (7 days), LAMA/LABA combination products if LAMA/LABA therapy is discontinued completely (Apply whichever mono component has the longest washout), Theophyllines (48 hours), Oral beta2-agonists (Long-acting [48 hours], short-acting [12 hours]), Inhaled short acting beta2-agonists (4 hours), Inhaled short-acting anticholinergics (4 hours), Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (4 hours), Any other investigational medication (30 days or within 5 drug half-lives [whichever is longer])
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulised Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulised therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.
* Previous participation in DB2113373 study: Subjects who have previously been assigned a subject number (enrolled) in GlaxoSmithKline study DB2113373.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2014-09-01; Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (11):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, San Antonio, Texas
- Bulgaria (7):
  - GSK Investigational Site, Dupnitsa
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Kyustendil
  - GSK Investigational Site, Montana
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
- Germany (5):
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Weyhe-Leeste, Lower Saxony
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (8):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szikszó
- Romania (6):
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
- Russia (9):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Sestroretsk
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yekaterinburg
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201211 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this randomized, double-blind, placebo-controlled parallel study, eligible participants received Umeclidinium/Vilanterol(UMEC/VI) 62.5/25 microgram(mcg) once daily(via Dry Powder Inhaler[DPI]) or matching placebo(1:1) for 12 weeks.The study consisted of Run-in Period(7-14 days), treatment period(12 weeks) and follow up period(7+-2 days).
Pre-assignment Details: A total of 627 participants who met eligibility criteria were screened; 498 participants were randomized and 496 comprised the Intent to Treat population.
Groups:
- Placebo: Participants with chronic obstructive pulmonary disease (COPD) received matching placebo via DPI once daily for 12 weeks. In addition, albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the run-in and double-blind treatment periods. Participants were followed up 7 days after the last dose of study medication.
- UMEC/VI 62.5/25 mcg: Participants with COPD received UMEC/VI 62.5/25mcg via DPI once daily for 12 weeks. In addition, albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the run-in and double-blind treatment periods. Participants were followed up 7 days after the last dose of study medication.
Period: Overall Study
Arm/Group | Placebo | UMEC/VI 62.5/25 mcg
Started | 248 | 248
Completed | 229 | 230
Not Completed | 19 | 18
Not completed — Adverse Event | 6 | 8
Not completed — Lack of Efficacy | 7 | 4
Not completed — Protocol deviation | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrew consent | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC/VI 62.5/25 mcg | Total
Number analyzed (Participants) | 248 | 248 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (8.23) | 64.1 (8.70) | 63.4 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 104 | 203
  Male | 149 | 144 | 293
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 4 | 7
  White - White/Caucasian/European | 245 | 244 | 489

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean St.George's Respiratory Questionnaire (SGRQ) Total Score at Day 84
Description: The SGRQ is a disease-specific questionnaire, self-completed by participants(par), used to evaluate the effect of UMEC/VI on health-related quality of life as compared to placebo in par with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Analysis was performed using mixed model repeated measures with covariates of Baseline (scores recorded prior to dosing on Day 1) SGRQ total score, centre group, smoking status, Day, treatment(trt), Day by Baseline interaction and Day by trt interaction, where Day is nominal. Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all par. randomized to trt. who received at least one dose of randomized study drug. Par. represents those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | UMEC/VI 62.5/25 mcg
Number analyzed (Participants) | 210 | 212
Score on scale | -2.12 (0.808) | -6.15 (0.803)
Statistical Analysis 1: Comparison: Placebo vs UMEC/VI 62.5/25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -4.03, 95% CI 2-sided [-6.28 to -1.79]

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 28, 56 and 84. Baseline is defined as the assessment taken pre-dose on Treatment Day 1. Trough FEV1 is defined as the FEV1 value obtained 24 hours after the previous morning's dosing. Change from Baseline at a particular visit was calculated as the trough FEV1 at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline , smoking status, center group, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | UMEC/VI 62.5/25 mcg
Number analyzed (Participants) | 224 | 227
Liter | 0.030 (0.0183) | 0.152 (0.0181)
Statistical Analysis 1: Comparison: Placebo vs UMEC/VI 62.5/25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 0.122, 95% CI 2-sided [0.071 to 0.172]

3. Secondary Outcome: Change From Baseline (BL) in Mean Number of Puffs of Rescue Medication Per Day Used Over Weeks 1-12
Description: Albuterol/salbutamol(A/S) was used as rescue medication and was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout treatment periods. The number of puffs of rescue medication (A/S) per day over the entire 12 week treatment period was recorded and analyzed. For rescue use, 'day' is referred as the period between one record of rescue use and the next. Total puffs of rescue for each day = number of salbutamol puffs + (2 x number of salbutamol nebules). Analysis performed using mixed model repeated measures with covariates of BL(mean number of total puffs over the duration from First Day; defined as Latest of [7 days before Visit 2 and day after Visit 1] to Last Day(defined as Day before Visit 2)), smoking status, centre group, four-week period, treatment and period by BL interaction. Change from BL used weeks 1-4, 5-8, and 9-12 as covariates in the model and the overall least squares mean change for weeks 1-12 is estimated.
Time Frame: Week 1 amd Week 12
Population: Intent-to-Treat (ITT) Population: all par. randomized to trt. who received at least one dose of randomized study drug. Par. represents all par. in the ITT population without missing covariate information and with at least one post BL measurement.
Measure: Least Squares Mean (Standard Error); unit: puffs per day
Groups:
- UMEC/VI 62.5/25mcg: Participants with COPD received UMEC/VI 62.5/25mcg via DPI once daily for 12 weeks. In addition, albuterol/salbutamol was provided to participants to use on an as-needed basis for relief of COPD symptoms throughout the run-in and double-blind treatment periods. Participants were followed up 7 days after the last dose of study medication.
Arm/Group | Placebo | UMEC/VI 62.5/25mcg
Number analyzed (Participants) | 247 | 244
puffs per day | -0.6 (0.13) | -1.4 (0.13)
Statistical Analysis 1: Comparison: Placebo vs UMEC/VI 62.5/25mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-1.1 to -0.4]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study drug untill follow-up (Follow-up is defined as up to Day 84 [-4 to +2 days]/Early withdrawal visit plus 7 days [± 2 days]).
Description: SAEs and non-serious AEs were collected in participants of the ITT population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Placebo | UMEC/VI 62.5/25mcg
Serious Adverse Events (participants affected / at risk) | 13/248 | 17/248
Other Adverse Events (participants affected / at risk) | 30/248 | 28/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=248) | UMEC/VI 62.5/25mcg (N=248)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pneumonia bacterial (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=248) | UMEC/VI 62.5/25mcg (N=248)
Headache (Nervous system disorders) | 16 | 16
Nasopharyngitis (Infections and infestations) | 16 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.